CLINICAL TRIAL: NCT03208140
Title: A Prospective, Multicenter Comparative Study of Laryngoscopic Vision With the TotalTrack Device Versus Indirect Laryngoscopy in Patients With an Uncomplicated Airway Scheduled for Surgery in the Context of Routine Anesthetic Practice
Brief Title: A Study of Laryngoscopic Vision With the TotalTrack Device Versus Indirect Laryngoscopy
Acronym: MULTITOTAL
Status: Completed | Type: Observational
Sponsor: Formacion Internacional para la Docencia e Investigación de la Vía Aérea (Other)
Responsible Party: Principal Investigator, pedro charco mora, Director, Formacion Internacional para la Docencia e Investigación de la Vía Aérea
Other Study IDs: HCV2017TTTK
Record Dates: First submitted 2017-06-10; First posted 2017-07-05 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Airway Obstruction; Difficult Intubation
Keywords: intubation to supraglottic devices; intubation device; laryngeal vision; success intubation; videolaryngoscope; direct intubation
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of the airway forms part of routine anesthetic practice. However, the predictions referred to intubation or ventilation difficulties are usually inconclusive. In effect, the failure rate in predicting such difficulties exceeds 60%. In this scenario it is not possible to know whether a given patient will be difficult to intubate and ventilate. These are referred to as non-intubate and non-ventilate cases with a high risk of severe neurological complications and even death due to hypoxemia. According to all the clinical guides, the solution in such cases usually involves the use of supraglottic devices that rescue oxygenation through effective ventilation.

In the event of ventilation failure with a supraglottic device, it is currently not possible to know whether the device is correctly positioned, unless some other instrument such as a flexible fiberscope is used to visualize the anatomy beyond the ventilation device.

The TotalTrack is a new device with all the characteristics of a supraglottic device that moreover includes a camera at the tip, allowing us to confirm anatomical positioning with respect to the glottic structures. This device also allows intubation under indirect visualization of the glottis, thus adding the possibility of definitive patient lung isolation.

The primary objective of this study is to determine the capacity to visualize the glottic structures through the camera of the TotalTrack device, compared with glottic visualization afforded by indirect laryngoscopy in the same patient. The Cormack-Lehane scale and percentage of glottic opening (POGO) are used for this purpose.

The secondary objectives comprise assessment of the ventilation, intubation and TotalTrack device withdrawal times. The hemodynamic changes associated to both techniques during intubation and TotalTrack device withdrawal are also evaluated. Minimum patient oxygenation throughout the procedure is assessed. The sealing and ventilation pressures during operation of the TotalTrack device are recorded. Likewise, an analysis is made of the number of placement attempts, visualization improvement maneuvers, and minor complications associated to the use of the TotalTrack device (presence of blood upon withdrawal or pharyngeal pain), with their degree of severity.

DETAILED DESCRIPTION:
The study hypothesis is that the new TTK device improves laryngoscopic visualization compared with direct laryngoscopy, thereby facilitating orotracheal intubation success.

The null hypothesis is that the new TTK device does not improve visualization of the glottic structures, the intubation conditions, or intubation success compared with direct laryngoscopy.

3. Objectives 3.1 Primary objective To determine whether the new TTK device improves laryngoscopic visualization as determined by the Cormack-Lehane scale and percentage of glottic opening (POGO), versus conventional laryngoscopy.

3.2 Secondary objectives

1. To assess intubation success, the laryngoscopy and intubation times, sealing pressure and subjective difficulty with the TTK intubation device.
2. To evaluate the hemodynamic impact, oxygenation and complications associated to the use of both intubation techniques.

4. Methodology 4.1 Type of study A prospective, multicenter, comparative observational study has been designed.

4.2 The study will begin following approval by the Clinical Research Ethics Committees of the participating hospitals, and will have an estimated duration of 9 months.

4.3 Study population The study will involve patients scheduled for surgery and requiring orotracheal intubation as routine practice.

According to the literature, the fibroscopic intubation success rate with other supraglottic devices is close to 98%, versus 95-98% in the case of direct laryngoscopy. Considering a 95% confidence interval and a study precision of 80%, the required sample size is 102 patients. A total of 30 patients will be enrolled per center in order to compensate for possible losses during follow-up.

4.4 Inclusion criteria Patients with ASA score I-III Age > 18 years Signing of the informed consent document

4.5. Exclusion criteria Age < 18 years Pregnant or breast-feeding women Patients with known difficult airways Patients requiring rapid sequence intubation

4.6 Study withdrawal criteria Patients who after inclusion in the study fail to comply with the protocol due to medical reasons, or who withdraw consent.

4. 7 Study protocol A prospective, multicenter, observational study has been designed, involving patients scheduled for surgery of any kind and requiring tracheal intubation, following the obtainment of informed consent. The study will include ASA I-III patients over 18 years of age. Individuals requiring rapid sequence intubation or diagnosed with difficult airways will be excluded.

Demographic data will be collected before anesthesia (age, gender, body mass index and ASA score), with evaluation of the airway (Mallampati score, thyroid-chin and sternum-chin distances, interincisal distance, upper lip bite test, neck flexion, dental prostheses, obstructive sleep apnea syndrome, presence of a beard and neck perimeter) and history of laryngoscopic procedures (if any). The patients also will be questioned about past neck irradiation, neck or ENT surgery and lingual tonsil hypertrophy, in order to predict supraglottic device management difficulties.

With the patient in the pre-operating room, a peripheral venous line will be prepared and premedication will be administered according to routine anesthetic practice.

Once in the operating room, standard monitoring will be carried out, with peripheral O2 saturation (SpO2) pulseoximeter, noninvasive arterial pressure (NIAP) and electrocardiography (ECG). The depth of hypnosis should be evaluated based on the bispectral index (BIS)(or through entropy monitoring), with the assessment of neuromuscular relaxation through train of four (TOF) monitoring.

Correct patient oxygenation will be performed during 3-5 minutes, with an inspiratory oxygen fraction of 100% using a correctly sealed face mask, with the aim of achieving an end-tidal O2 level of over 90% (ETO2 > 0.9). Following the above, anesthesia induction will be carried out with fentanyl (1-2 µg kg-1), propofol (2-3 mg kg-1) and rocuronium (0.6 mg kg-1). Endotracheal intubation will be performed when TOF = 0. Conventional laryngoscopy will be carried out using a Macintosh blade in all patients, recording the exploration times and the best laryngeal visualization achieved (using the Cormack-Lehane scale and percentage of glottic opening [POGO]) with or without BURP (backward, upward and rightward pressure on the thyroid cartilage) maneuvering. The best laryngeal vision achieved after these maneuvers will be recorded. The TotalTrack (TTK) video laryngeal mask will then be placed.

Prior to intubation with this new device, the investigators will measure the TTK sealing pressure, setting the respirator to manual mode, closing the expiratory valve to 40 cmH2O, and adjusting the fresh gas flow to 3 litres. The pressure at which audible leakage occurs will be measured. If the pressure exceeds 40 cmH2O, the test will be considered over, and this latter value will be recorded as the TTK sealing pressure (> 40 cmH2O).

Lastly, intubation will be carried out with an endotracheal tube half a grade less than the maximum recommended by the manufacturer of the TTK.

During both direct laryngoscopy and after placement of the TTK, the best laryngoscopic vision achieved will be recorded, based on the Cormack-Lehane scale and POGO, together with the laryngoscopy and intubation times. The laryngoscopy time is defined as the time elapsed from insertion of the laryngoscope or study device through the teeth to best vision of the glottis. The intubation time in turn is defined as the time elapsed from collapse of the endotracheal tube cuff to definitive positioning of the instrument beyond the vocal cords (insertion mark on the tube), following capnographic confirmation of correct intubation. If correct positioning is not achieved, the maneuver will be repeated, recording the time from collapse of the cuff in the esophagus to correct positioning of the endotracheal tube. The times will be recorded as accurately as possible. The use of a chronometer is advised.

Data will be collected referred to heart rate, blood pressure (systolic / diastolic) and BIS / entropy monitoring at the following times:

1. Before the induction of anesthesia (baseline value)
2. Two minutes after the induction of anesthesia (post-induction baseline value)
3. Immediately after direct laryngoscopy (post-direct laryngoscopy stress response)
4. Before insertion of the TTK (post-direct laryngoscopy baseline value)
5. Immediately after insertion of the TTK (post-TTK stress response)
6. After tracheal intubation (post-intubation stress response)

The BIS will be within anesthetic values at all times. If necessary, additional hypnotic drug doses (propofol) will be administered (to be reflected in the total administered dosage).

Evaluation of the subjective technical difficulty of the new device will be based on a numerical scale from 1-10 (1 = very easy, 10 - insertion impossible).

Other data to be recorded for assessing the difficulties of the two techniques are the need for repositioning of the TTK, external laryngeal manipulation maneuvers (BURP, lateralization of the neck), the use of assists in intubation, and the number of attempts required to secure orotracheal intubation.

The following complications will be documented: esophageal intubation; trauma of the mouth, lips, tongue or teeth; presence of blood in the device; throat pain and dysphonia (in the post-anesthesia recovery unit and 24 hours after surgery).

5. Statistical analysis A descriptive analysis will be made of all the variables, including the demographic data, predictors of difficult intubation, number of insertion and intubation attempts, and the TTK intubation and withdrawal times. Continuous variables will be reported as the mean and standard error, while categorical variables will be reported as frequency and percentage. The chi-squared test will be used to compare categorical variables, while quantitative variables will be contrasted using the Student t-test. The data will be analyzed using the Statistical Package for the Social Sciences (SPSS, Chicago, IL, USA), version 20.0.

7. Strengths of the study If the study is successfully completed, the anesthesiologist will have a new tool for orotracheal intubation that may minimize complications in the case of difficult airways - thereby reducing healthcare resource utilization and the length of hospital stay.

The use of this device in the management of expected or unexpected difficult airways could avoid important postoperative complications associated to such difficulties. In future, increased experience and a larger number of patients could consolidate the TTK in an important position in the difficult airway management algorithms.

8. Expected impact

If the study hypothesis is correct, the benefits of improvement in the intubation technique include:

* A lesser risk of complications derived from hypoxemia, including irreversible brain damage and death.
* Early discharge from the post-anesthesia recovery unit (PARU).
* Early discharge from hospital.
* Significant reduction of healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA score I-III
* Age > 18 years
* Signing of the informed consent document

Exclusion Criteria:

* Age < 18 years
* Pregnant or breast-feeding women
* Patients with known difficult airways
* Patients requiring rapid sequence intubation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who after inclusion in the study fail to comply with the protocol due to medical reasons, or who withdraw consent.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
To determine whether the new TTK device improves laryngoscopic visualization | Time of Orotracheal intubation (up to 1 hour)
  To determine whether the new TTK device improves laryngoscopic visualization as determined by the Cormack-Lehane, versus conventional laryngoscopy.

SECONDARY OUTCOMES:
To assess intubation success, | Time of Orotracheal intubation (up to 1 hour)
  Record number of the total intubation success
To assess the laryngoscopy times | Time of Orotracheal intubation (up to 1 hour)
  Record the times in seconds of the best glottic vision
To assess the intubation times | Time of Orotracheal intubation (up to 1 hour)
  Record the times in seconds of the pass the tube for glottic inlet
To determinate pressure sealing of the totaltrack device (laryngeal mask) | post totaltrack introduction and correct pressure ventilation (until 10 minutes)
  Record the pressure Totaltrack's (mmHg) mask determinate with manometer pressure
To determinate hemodynamic parameters during totaltrack insertion | Time postTotaltrack insertion (up to 10 minutes)
  Record arterial pressure (mmHg) during direct laryngoscopy
To determinate hemodynamic parameters during direct laryngoscopy | Time post direct laryngoscopy (up to 10 minutes)
  Record arterial pressure (mmHg) during direct laryngoscopy
To determinate hemodynamic parameters during intubation | Time postOrotracheal intubation (up to 10 minutes)
  Record arterial pressure (mmHg) during intubation
To determinate complication of the technical intubation | immediately postintubation and 24 hours later (up to 24 hours)
  Record throat pain (analogic visual scale 1=no pain to10= maximal pain)and dysphonia (light-moderate-severe)in immediate postoperatory and next day

CONTACTS AND LOCATIONS:
Overall Officials: pedro Charco-Mora, MD, PhD, Study Chair — Formacion Internacional para la Docencia e Investigación de la Vía Aérea
Locations (2):
- Spain (2):
  - Pedro Charco Mora, Valencia
  - Pedro Charco-Mora, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ott T, Barth A, Kriege M, Jahn-Eimermacher A, Piepho T, Noppens RR. The novel video-assisted intubating laryngeal mask Totaltrack compared to the intubating laryngeal mask Fastrach - a controlled randomized manikin study. Acta Anaesthesiol Scand. 2017 Apr;61(4):381-389. doi: 10.1111/aas.12872. PMID 28251605
- [Background] Langenstein H, Moller F. [The importance of the laryngeal mask in the difficult intubation and early experience with the intubating laryngeal mask airway--ILMA--Fastrach]. Anasthesiol Intensivmed Notfallmed Schmerzther. 1998 Dec;33(12):771-80. doi: 10.1055/s-2007-994852. German. PMID 9893911
- [Background] Izquierdo-Gonzalez B, Gomez-Rios MA, Freire-Vila E. Use of the TotalTrack VLM for emergent endotracheal intubation in predicted difficult airway with obstruction by expanding space-occupying lesions and reduced interincisor opening. Rev Esp Anestesiol Reanim. 2017 Aug-Sep;64(7):415-418. doi: 10.1016/j.redar.2017.01.004. Epub 2017 Mar 2. English, Spanish. PMID 28262247
- [Background] Gaszynski T. TotalTrack video intubating laryngeal mask in super-obese patients - series of cases. Ther Clin Risk Manag. 2016 Mar 2;12:335-8. doi: 10.2147/TCRM.S95695. eCollection 2016. PMID 27042078
- [Background] Aleksandrowicz D, Gaszynski T. Airway Management with Cervical Spine Immobilisation: A Comparison between the Macintosh Laryngoscope, Truview Evo2, and Totaltrack VLM Used by Novices--A Manikin Study. Biomed Res Int. 2016;2016:1297527. doi: 10.1155/2016/1297527. Epub 2016 Feb 29. PMID 27034926
- [Background] Gomez-Rios MA, Freire-Vila E, Vizcaino-Martinez L, Estevez-Gonzalez E. The Totaltrack: an initial evaluation. Br J Anaesth. 2015 Nov;115(5):799-800. doi: 10.1093/bja/aev336. No abstract available. PMID 26475813
- [Background] Acha Gandarias P. [Advances in airway management: The future is here]. Rev Esp Anestesiol Reanim. 2016 Jan;63(1):1-2. doi: 10.1016/j.redar.2015.10.006. Epub 2015 Nov 28. No abstract available. Spanish. PMID 26642950